CLINICAL TRIAL: NCT05137028
Title: Effects of Otago Exercise on Balance and Mobility in Patient With Total Knee Replacement
Brief Title: Otago Exercise in Patient With Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/01042 Allena Javed
Record Dates: First submitted 2021-11-18; First posted 2021-11-30 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Total Knee Replacement
Keywords: Balance training; Total knee replacement; Otago exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Otago Exercise (Experimental): Otago Exercise Group
  Interventions: Other: Otago Exercise

INTERVENTIONS:
Other: Otago Exercise — Otago exercise protocol
  Strengthening exercise:
  Resistance exercise for knee flexors, knee extensors, hip abductor, ankle dorsiflexors, ankle planterflexors
  Balance exercise:
  knee bending, backward walking, walking and turning around, sideway walking, tendem stance, tendem walking, one leg stand, heel walking, toe walking, heel to toe walking, sit to stand, stair walking

SUMMARY:
To determine the effect of Otago exercise in Total Knee Replacement

DETAILED DESCRIPTION:
Degenerative knee arthritis is one of the most common diseases in the elderly population. Age is the strongest risk factor for osteoarthritis. The 2010 Global Burden of Disease Study reports that the burden of musculoskeletal disorders is much larger than estimated in previous assessments and accounts for 6.8% of daily worldwide. An estimated 10% to 15% of all adults aged over 60 have some degree of OA. In Pakistan, 3.6% in rural and 3.1-4.6% in urban parts of Pakistan were found diagnosed by knee OA.

When conservative treatments fail to control the symptoms, joint replacement is performed. Specifically, more than 1 million surgeries are performed every year in the United States (US) alone, with a total expenditure close to 13.7 billion and 28.5 billion US dollars for the hips and knees, respectively. The demand is expected to increase by approximately 4 time by the year 2030 annually more than 4000 joint have been replaced in Pakistan." Overall, the progress of patients after joint replacement is satisfactory. Nevertheless, a substantial number may present with functional and balance limitations, even 1 year after surgery.

A cross sectional study reported that a Home-based balance and strength exercises (OEP) benefited older fallers with OA and gait and balance disorders by improving postural control. Another study has been done which suggested that elderly people who performed the OEP showed an increase in balance, muscle strength, and a decrease in both fall percentage and fall frequency. Evidence has recommended that, the OEP was more effective improving functional balance, muscle strength and physical health.

A cross sectional study was conducted to evaluate the influence of specific balance-targeted training on the overall state of balance in older adults undergoing TKR. They concluded that the additional balance training program improved balance performance to a higher extent than a control group.

After surgery, pain and stiffness are remarkably relieved, but functional and proprioceptive deficits, including limitation of lower limb mobility, difficulties in walking, and alterations instability and balance may remain. However, the effect of Otago exercise on balance are present in literature but the evidence for their influence in patients with TKR is narrow. So aim of this study to identify the possible role of Otago exercise program in particular population (TKR) and the prognosis in balance and Gait with this protocol in patients undergoing TKR.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Participants who undergo unilateral cemented knee replacement due to arthritis

Exclusion Criteria:

* Uncontrolled Hypertension
* Lower extremity impairment that can limit the patient's function
* Patient with neurological and cognitive impairment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
The Functional Reach test | 24 weeks
  The Functional Reach Test is a single item test developed as a quick screen for balance problems in older adults. It ranges 6-10 inches greater than 10 inches indicate low risk of fall as lower than 6 inches has higher risk of fall.
Timed Up and Go (TUG) Test | 24 weeks
  Measure of function with correlates to balance and fall risk. Less than 10 seconds for this task means normal while greater seconds mean higher risk of fall
Single leg Stance (SLS) Test | 24 weeks
  The Single leg Stance (SLS) Test is used to assess static postural and balance control. Single leg stance more than 10 seconds is normal. Less than 5 seconds indicate higher risk of fall.
Stair Climbing Test | 24 weeks
  Stair climbing test is used to assess Functional strength, balance and agility through ascending and descending a set number of steps. 5 minutes for 9 step of stairs means normal while more than 5 minutes for 9 step of stairs indicate risk of fall.
Balance and Gait App | 24 weeks
  This app will use to assess the balance and gait. It has 4 competent 2 for static and 2 for dynamic. For static patient will stand for eyes open and close, and for dynamic patient will walk for 3 meter with and without head movement. Maximum time for each task is 30 seconds. For dynamic balance the average range for this age groups is 60-67 lower than this indicate higher risk of fall.
Numerical Pain Rating Scale | 24 weeks
  Numeric Pain Rating Scale NPRS measure of the intensity of pain. Numerical pain rating scores is 0-10. 0 means no pain while 10 means worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Study Chair — Riphah International University
Locations (1):
- Umer Bashir Hospital, Lalamusa, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No